CLINICAL TRIAL: NCT05238779
Title: An Integrative Model for Palliative Care in End-Stage Liver Disease
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20023178
Record Dates: First submitted 2022-02-07; First posted 2022-02-14 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: End Stage Liver DIsease
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- End Stage Liver Disease (ESLD): Patients with ESLD
  Interventions: Other: Standard of care including palliative care

INTERVENTIONS:
Other: Standard of care including palliative care — Usual care includes laboratory evaluations, imaging, and certain procedures and medications. In some cases of patients undergoing transplant evaluation, usual care will also include multiple visits with members of the liver transplant team. A palliative care consult will also be part of standard of care. The primary goal of the palliative care consult is not to arrange hospice (though that can be done in appropriate situations) but to identify and try to address the impacts of the disease and its symptoms on patient's life.

SUMMARY:
The purpose of this research study is to understand the impact of palliative care in ESLD on quality of life, emergency room or hospital visits, and on care provider burden, and to work to develop the best way to provide palliative care in ESLD.

DETAILED DESCRIPTION:
Patients with end-stage liver disease (ESLD) have multiple symptoms that impact their quality of life and result in more emergency room and hospital visits. Palliative care is a medical model that can help alleviate pain and suffering and reduce need for urgent medical care and can do so while continuing other appropriate medical care. While palliative care consults are used in those with ESLD, despite the pain and suffering that accompanies ESLD, palliative care is often used too little and too late.

ELIGIBILITY:
Inclusion Criteria:

Primary participant:

* admission for decompensated cirrhosis, age ≥ 18
* willingness to sign consent
* able to read and understand English
* presence of decompensated cirrhosis with portal hypertension (jaundice, ascites, HE, hepatohydrothorax, AKI, HRS and/or variceal bleeding) or HCC

Caregiver:

* identified as the primary caregiver of the participant
* age ≥ 18
* willingness to sign consent
* able to read and understand English

Exclusion Criteria:

Primary participant:

* prior liver transplant
* lack of capacity to provide informed consent (in the judgement of the investigator)
* already in receipt of palliative or hospice care
* those who are likely to receive a LT during the index admission

Caregiver:

• none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with ESLD and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Change in symptom intensity | Up to 60 days
  Edmonton Symptom Assessment System (ESAS) - participants rate the intensity of common symptoms on 0-10 scale with 0= no symptom and 10=worst symptom imaginable. Scores range from 0 to 90 with higher scores indicating worse symptoms.
Change in liver disease QOL | Up to 60 days
  Short-Form Liver Disease QOL - The SF-LDQOL includes 36 disease-targeted items representing nine domains: symptoms of liver disease, effects of liver disease, memory/concentration, sleep, hopelessness, distress, loneliness, stigma of liver disease and sexual problems. The minimum and maximum values of the scale are 0-100 with higher scores indicating better QOL.
Change in depression | Up to 60 days
  Patient Health Questionnaire 9 (PHQ-9) is a self-report instrument which assesses depression. Scores range from 0 to 27 with higher scores indicating worse depression.
Change in anxiety | Up to 60 days
  Generalized Anxiety Disorder 7-Item Scale (GAD-7) is a self-report instrument which assesses anxiety. Scores range from 0 to 21 with higher scores indicating greater anxiety.
Change in perform ordinary tasks | Up to 60 days
  The Karnofsky Performance Status will be used to assess participants ability to perform ordinary tasks. Scores range from 0 to 100 with higher scores indicating greater ability.
Change in caregiver burden | Up to 60 days
  The Zarit Burden Interview
Hospital readmissions and/or Emergency room (ER) visits | 60 days
  Number of participants with ER visits or who are readmitted to the hospital during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Joel Wedd, MD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No